CLINICAL TRIAL: NCT02779543
Title: Clinical Validation of New Commercial Sleep Monitoring Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1509016542
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea
Keywords: In lab sleep studies
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Fitbit (Active Comparator): Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non dominant hand when prepared for the sleep study by a technician. Subjects willing to wear more than one sleep monitoring device may be fitted with two different sleep monitoring devices, e.g., a Fitbit and a Jawbone UP or a Fitbit and a Microsoft Band. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Interventions: Device: Fitbit
- Jawbone UP (Active Comparator): Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non dominant hand when prepared for the sleep study by a technician. Subjects willing to wear more than one sleep monitoring device may be fitted with two different sleep monitoring devices, e.g., a Fitbit and a Jawbone UP or a Fitbit and a Microsoft Band. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Interventions: Device: Jawbone UP
- Microsoft Band (Active Comparator): Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non dominant hand when prepared for the sleep study by a technician. Subjects willing to wear more than one sleep monitoring device may be fitted with two different sleep monitoring devices, e.g., a Fitbit and a Jawbone UP or a Fitbit and a Microsoft Band. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Interventions: Device: Microsoft Band

INTERVENTIONS:
Device: Fitbit — Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non-dominant hand when prepared for the sleep study by a technician.
  Arms: Fitbit
Device: Jawbone UP — Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non-dominant hand when prepared for the sleep study by a technician.
  Arms: Jawbone UP
Device: Microsoft Band — Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non-dominant hand when prepared for the sleep study by a technician.
  Arms: Microsoft Band

SUMMARY:
This study seeks to validate three new commercial sleep monitoring devices: Fitbit, Jawbone UP, and Microsoft Band by comparison against concurrent polysomnography (PSG), which is considered the gold standard for sleep assessment. This research is being done because if proven to accurately analyze sleep,these devices may make conducting in-home sleep studies easier and more affordable in the future.

DETAILED DESCRIPTION:
This study seeks to validate three new commercial sleep monitoring devices: Fitbit, Jawbone UP, and Microsoft Band by comparison against concurrent polysomnography (PSG), considered the gold standard assessment for sleep physiology. The investigators emphasize here that the commercial sleep monitoring devices (Fitbit, Jawbone UP, and Microsoft Band) are used in addition to PSG and not in place of it. Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine. Willing subjects, after providing informed consent, will be fitted with one of the three aforementioned sleep monitoring devices (randomly assigned) on the wrist of their non-dominant hand when prepared for the sleep study by a technician. Subjects willing to wear more than one sleep monitoring device may be fitted with two different sleep monitoring devices, e.g., a Fitbit and a Jawbone UP or a Fitbit and a Microsoft Band. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study. Data will be transferred from the sleep monitoring device(s) for later statistical analysis and comparison with scored polysomnogram. Device(s) will be cleaned (using antiseptic wipes), reset,recharged, and otherwise prepared for reuse.

ELIGIBILITY:
Inclusion Criteria:

* Attending a regularly scheduled overnight polysomnography (PSG) sleep study at the Weill Cornell Medical College Center for Sleep Medicine.

Exclusion Criteria:

* Not attending a regularly scheduled overnight polysomnography (PSG) sleep study at the Weill Cornell Medical College Center for Sleep Medicine.
* Under 18 or over 80 years old.
* Pregnancy
* Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Krieger, M.D., M.P.H, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine Center for Sleep Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fitbit Charge 2: Willing subjects, after providing informed consent, will be fitted with Fitbit Charge 2 on the wrist of their non dominant hand when prepared for the sleep study by a technician. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Fitbit: Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine.
- Microsoft Band 2: Willing subjects, after providing informed consent, will be fitted with Microsoft Band 2 on the wrist of their non dominant hand when prepared for the sleep study by a technician. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Microsoft Band 2: Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine.
Period: Overall Study
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This arm was dropped due to cost restrictions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fitbit Charge 2 | Microsoft Band 2 | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 75 | 138
  >=65 years | 37 | 25 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 81
  Male | 58 | 61 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 100 | 100 | 200
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time as Measured by Fitbit Charge2 or Microsoft Band2.
Description: Statistical analysis will examine agreement levels of sleep metrics such as Total Sleep Time (TST).
Time Frame: 1 night, approximately 9 hours.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Microsoft Band 2: Willing subjects, after providing informed consent, will be fitted with Microsoft Band 2 on the wrist of their non dominant hand when prepared for the sleep study by a technician. Sleep monitoring device(s) will be removed from the subject's wrist in the morning at the conclusion of the sleep study.
  Fitbit: Subjects will be recruited from those patients attending a regularly scheduled overnight PSG sleep study at the Weill Cornell Medical College Center for Sleep Medicine.
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
Number analyzed (Participants) | 100 | 100
minutes | 437.0 (80.6) | 394.9 (105.8)
Statistical Analysis 1: Comparison: Fitbit Charge 2 vs Microsoft Band 2; Test type: Equivalence — this trial compared the 2 devices to the polysomnography, which is the gold standard; p < 0.001, ANOVA; Mean value = 368.3 — compared to gold standard

2. Secondary Outcome: Sleep Onset Latency as Measured by Fitbit Charge2 or Microsoft Band2.
Description: Statistical analysis will examine agreement levels of sleep metrics such as Sleep Onset Latency (SOL).
Time Frame: 1 night, approximately 9 hours.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
Number analyzed (Participants) | 100 | 100
minutes | 8.8 (13.7) | 26.2 (30.5)
Statistical Analysis 1: Comparison: Fitbit Charge 2 vs Microsoft Band 2; Test type: Equivalence — This trial compared those 2 devices with the gold standard (polysomnography); p < 0.001, ANOVA; Mean value = 13.9 — compared to gold standard

3. Secondary Outcome: Wake Time After Sleep Onset as Measured by Fitbit Charge2 or Microsoft Band2.
Description: Statistical analysis will examine agreement levels of sleep metrics such as Wake After Sleep Onset (WASO)
Time Frame: 1 night, approximately 9 hours.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
Number analyzed (Participants) | 100 | 100
minutes | 30.3 (42.0) | 88.0 (71.7)
Statistical Analysis 1: Comparison: Fitbit Charge 2 vs Microsoft Band 2; Test type: Equivalence — This trial compared those 2 devices with the gold standard (polysomnography); p < 0.001, ANOVA; Mean value = 106 — compared to gold standard

4. Secondary Outcome: Sleep Efficiency as Measured by Fitbit Charge2 or Microsoft Band2.
Description: Statistical analysis will examine agreement levels of sleep metrics such as Sleep Efficiency (SE)
Time Frame: 1 night, approximately 9 hours.
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
Number analyzed (Participants) | 100 | 100
percentage of sleep efficiency | 93.4 (9.6) | 82.1 (15.5)
Statistical Analysis 1: Comparison: Fitbit Charge 2 vs Microsoft Band 2; Test type: Equivalence — This trial compared those 2 devices with the gold standard (polysomnography); p < 0.001, ANOVA; Mean value = 74.3 — compared to gold standard

ADVERSE EVENTS:
Time Frame: 1 day - the day after the recording night when the device was worn
Arm/Group | Fitbit Charge 2 | Microsoft Band 2
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol, Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT02779543/Prot_SAP_000.pdf